CLINICAL TRIAL: NCT00121667
Title: "A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Trial to Evaluate the Efficacy and Safety of BMS-477118 in Combination With Metformin in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Alone"
Brief Title: Study Assessing Saxagliptin Treatment In Type 2 Diabetic Subjects Who Are Not Controlled With Metformin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-014
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Results first posted 2011-04-08 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Saxagliptin + Metformin (A) (Experimental): Pioglitazone 15-45 mg (as needed for rescue)
  Interventions: Drug: Saxagliptin + Metformin; Drug: Pioglitazone
- Saxagliptin + Metformin (B) (Experimental): Pioglitazone 15-45 mg (as needed for rescue)
  Interventions: Drug: Saxagliptin + Metformin; Drug: Pioglitazone
- Saxagliptin + Metformin (C) (Experimental): Pioglitazone 15-45 mg (as needed for rescue)
  Interventions: Drug: Saxagliptin + Metformin; Drug: Pioglitazone
- Placebo+ Metformin (D) (Placebo Comparator): Pioglitazone 15-45 mg (as needed for rescue)
  Interventions: Drug: Placebo + Metformin; Drug: Pioglitazone

INTERVENTIONS:
Drug: Saxagliptin + Metformin — Tablets, Oral, 2.5 mg Saxagliptin (plus flexible metformin dose), Once daily (24 weeks ST, 42 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin + Metformin (A)
Drug: Saxagliptin + Metformin — Tablets, Oral, 5 mg Saxagliptin (plus flexible metformin dose), Once daily (24 weeks ST, 42 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin + Metformin (B)
Drug: Saxagliptin + Metformin — Tablets, Oral, 10 mg Saxagliptin (plus flexible metformin dose), Once daily (24 weeks ST, 42 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin + Metformin (C)
Drug: Placebo + Metformin — Tablets, Oral, 0 mg, Once daily (24 weeks ST, 42 months LT)
  Arms: Placebo+ Metformin (D)
Drug: Pioglitazone — Tablets, Oral, 15 - 45 mg (as needed for rescue)

SUMMARY:
The purpose of this clinical research study is to learn whether Saxagliptin added to Metformin therapy is more effective than Metformin alone as a treatment for type 2 diabetic subjects who are not sufficiently controlled with Metformin alone

DETAILED DESCRIPTION:
All subjects will participate in a lead-in period, and qualifying subjects will continue into a short-term randomized treatment period. Subjects who complete the short-term period will be eligible to enter the long term extension period. Also, subjects in the short-term period who have an elevated blood sugar that requires additional medication for blood sugar control will be eligible to enter the long-term treatment extension period where they will receive pioglitizone added onto their blinded study medication

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus requiring treatment with at least 1500 mg but not greater than 2550 mg of a maximum tolerated dose of Metformin therapy for at least 8 weeks prior to screening.
* HbA1c >= 7.0% and <= 10.0 %
* Body mass index <= 40 kg/m2
* Fasting C-peptide >= 1 ng/dL

Exclusion Criteria:

* Symptomatic poorly controlled diabetes
* Recent cardiac or cerebrovascular event
* Serum creatinine >= 1.5 mg/dL for males and >= 1.4 mg/dL for females

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1462 (Actual)
Dates: Start 2005-08; Primary Completion 2006-10 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (152):
- United States (95):
  - Local Institution, Anniston, Alabama
  - Local Institution, Birmingham, Alabama
  - Local Institution, Calera, Alabama
  - Local Institution, Haleyville, Alabama
  - Local Institution, Mesa, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution, Jonesboro, Arkansas
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Sherwood, Arkansas
  - Local Institution, Encino, California
  - Local Institution, Fountain Valley, California
  - Local Institution, Fresno, California
  - Local Institution, Los Angeles, California
  - Local Institution, Mission Viejo, California
  - Local Institution, Northridge, California
  - Local Institution, Orange, California
  - Local Institution, Roseville, California
  - Local Institution, Sacramento, California
  - Local Institution, Spring Valley, California
  - Local Institution, Tustin, California
  - Local Institution, Castle Rock, Colorado
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Denver, Colorado
  - Local Institution, Golden, Colorado
  - Local Institution, Loveland, Colorado
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Chipley, Florida
  - Local Institution, Cocoa Beach, Florida
  - Local Institution, Coral Gables, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Kissimmee, Florida
  - Local Institution, Marianna, Florida
  - Local Institution, Miami, Florida
  - Local Institution, New Port Richey, Florida
  - Local Institution, Ocala, Florida
  - Local Institution, Tallahassee, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Decatur, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Vernon Hills, Illinois
  - Local Institution, Elkhart, Indiana
  - Local Institution, Lafayette, Indiana
  - Local Institution, Iowa City, Iowa
  - Local Institution, Waterloo, Iowa
  - Local Institution, Topeka, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Munfordville, Kentucky
  - Local Institution, New Orleans, Louisiana
  - Local Institution, West Monroe, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Chester, Maryland
  - Local Institution, Prince Frederick, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Kalispell, Montana
  - Local Institution, Omaha, Nebraska
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Toms River, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Greensboro, North Carolina
  - Local Institution, Morehead City, North Carolina
  - Local Institution, Salisbury, North Carolina
  - Local Institution, Sparta, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Athens, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Lyndhurst, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Eugene, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Carlisle, Pennsylvania
  - Local Institution, Langhorne, Pennsylvania
  - Local Institution, Levittown, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Duncan, South Carolina
  - Local Institution, Bristol, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Bryan, Texas
  - Local Institution, Carrollton, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Temple, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Hampton, Virginia
  - Local Institution, Virginia Beach, Virginia
  - Local Institution, Olympia, Washington
  - Local Institution, Spokane, Washington
- Argentina (4):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
- Australia (8):
  - Local Institution, Sydney, New South Wales
  - Local Institution, Woollongong, New South Wales
  - Local Institution, Brisbane, Queensland
  - Local Institution, Kippa-Ring, Queensland
  - Local Institution, Meadowbrook, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Woodville South, South Australia
  - Local Institution, Perth, Western Australia
- Brazil (6):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Belém, Pará
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Campinas, São Paulo
  - Local Institution, Marília, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (23):
  - Local Institution, Calgary, Alberta
  - Local Institution, Coquitlam, British Columbia
  - Local Institution, Kelowna, British Columbia
  - Local Institution, Surrey, British Columbia
  - Local Institution, Brandon, Manitoba
  - Local Institution, Portage la Prairie, Manitoba
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, Mount Pearl, Newfoundland and Labrador
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Aylmer, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Oakville, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Thornhill, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Woodstock, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Drummondville, Quebec
  - Local Institution, Fleurimont, Quebec
  - Local Institution, Longueuil, Quebec
  - Local Institution, Saint-Léonard, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Mexico (8):
  - Local Institution, Durango, Durango
  - Local Institution, Celaya, Guanajuato
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Distrito Federal, Mexico City
  - Local Institution, Morelia, Michioacan
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Hermosillo, Sonora
  - Local Institution, Mérida, Yucatán
- Puerto Rico (4):
  - Local Institution, Carolina
  - Local Institution, Ponce
  - Local Institution, Rio Pieoras
  - Local Institution, San Juan
- Taiwan (3):
  - Local Institution, Hualien City
  - Local Institution, Taichung
  - Local Institution, Taipei

REFERENCES:
- [Background] DeFronzo RA, Hissa MN, Garber AJ, Luiz Gross J, Yuyan Duan R, Ravichandran S, Chen RS; Saxagliptin 014 Study Group. The efficacy and safety of saxagliptin when added to metformin therapy in patients with inadequately controlled type 2 diabetes with metformin alone. Diabetes Care. 2009 Sep;32(9):1649-55. doi: 10.2337/dc08-1984. Epub 2009 May 28. PMID 19478198
- [Derived] Bailey CJ, Del Prato S, Wei C, Reyner D, Saraiva G. Durability of glycaemic control with dapagliflozin, an SGLT2 inhibitor, compared with saxagliptin, a DPP4 inhibitor, in patients with inadequately controlled type 2 diabetes. Diabetes Obes Metab. 2019 Nov;21(11):2564-2569. doi: 10.1111/dom.13841. Epub 2019 Aug 26. PMID 31364269
- [Derived] Perl S, Cook W, Wei C, Iqbal N, Hirshberg B. Saxagliptin Efficacy and Safety in Patients With Type 2 Diabetes and Moderate Renal Impairment. Diabetes Ther. 2016 Sep;7(3):527-35. doi: 10.1007/s13300-016-0184-9. Epub 2016 Jul 11. PMID 27402391
- [Derived] Bonora E, Bryzinski B, Hirshberg B, Cook W. A post hoc analysis of saxagliptin efficacy and safety in patients with type 2 diabetes stratified by UKPDS 10-year cardiovascular risk score. Nutr Metab Cardiovasc Dis. 2016 May;26(5):374-9. doi: 10.1016/j.numecd.2015.11.004. Epub 2015 Dec 1. PMID 27033025
- [Derived] Rosenstock J, Gross JL, Aguilar-Salinas C, Hissa M, Berglind N, Ravichandran S, Fleming D. Long-term 4-year safety of saxagliptin in drug-naive and metformin-treated patients with Type 2 diabetes. Diabet Med. 2013 Dec;30(12):1472-6. doi: 10.1111/dme.12267. Epub 2013 Jul 19. PMID 23802840
- [Derived] Karyekar CS, Frederich R, Ravichandran S. Clinically relevant reductions in HbA1c without hypoglycaemia: results across four studies of saxagliptin. Int J Clin Pract. 2013 Aug;67(8):759-67. doi: 10.1111/ijcp.12212. Epub 2013 Jun 24. PMID 23795975
- [Derived] Karyekar C, Donovan M, Allen E, Fleming D, Ravichandran S, Chen R. Efficacy and safety of saxagliptin combination therapy in US patients with type 2 diabetes. Postgrad Med. 2011 Jul;123(4):63-70. doi: 10.3810/pgm.2011.07.2305. PMID 21680990

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1462 participants were enrolled, and 787 entered the lead-in period. 45 discontinued the during the lead-in period. 19 subjects no longer met study criteria, 10 subjects withdrew consent, and 2 subjects were randomized but not treated.
Groups:
- Saxagliptin 2.5 mg + Metformin: Tablets, Oral, 2.5 mg Saxagliptin (plus flexible metformin dose), Once daily (24 weeks ST, 42 months LT); Pioglitazone 15-45 mg (as needed for rescue).
- Saxagliptin 5 mg + Metformin: Tablets, Oral, 5 mg Saxagliptin (plus flexible metformin dose), Once daily (24 weeks ST, 42 months LT); Pioglitazone 15-45 mg (as needed for rescue).
- Saxagliptin 10 mg + Metformin: Tablets, Oral, 10 mg Saxagliptin (plus flexible metformin dose), Once daily (24 weeks ST, 42 months LT); Pioglitazone 15-45 mg (as needed for rescue).
- Placebo+ Metformin: Tablets, Oral, 0 mg, Once daily (24 weeks ST, 42 months LT); Pioglitazone 15-45 mg (as needed for rescue).
Period: Short Term (ST) Period
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Started | 192 | 191 | 181 | 179
Completed | 148 | 143 | 140 | 112
Not Completed | 44 | 48 | 41 | 67
Not completed — Lack of Efficacy | 25 | 22 | 27 | 44
Not completed — Subject Withdrew Consent | 8 | 13 | 4 | 11
Not completed — Adverse Event | 5 | 6 | 5 | 3
Not completed — Lost to Follow-up | 3 | 4 | 4 | 3
Not completed — Poor / Non-compliance | 0 | 1 | 1 | 2
Not completed — Subject No Longer Meets Study Criteria | 0 | 2 | 0 | 2
Not completed — Other Reason | 3 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1
Period: Short Term (ST) + Long Term (LT) Period
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Started | 192 | 191 | 181 | 179
Completed Study Without Being Rescued | 14 | 18 | 23 | 7
Completed | 64 | 58 | 68 | 39
Not Completed | 128 | 133 | 113 | 140
Not completed — Lack of Efficacy | 54 | 51 | 42 | 65
Not completed — Subject Withdrew Consent | 38 | 34 | 26 | 30
Not completed — Adverse Event | 12 | 18 | 13 | 10
Not completed — Lost to Follow-up | 11 | 11 | 13 | 16
Not completed — Other Reason | 5 | 7 | 6 | 3
Not completed — Subject No Longer Meets Study Criteria | 3 | 6 | 5 | 9
Not completed — Poor / Non-compliance | 3 | 5 | 8 | 4
Not completed — Pregnancy | 1 | 1 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin | Total
Number analyzed (Participants) | 192 | 191 | 181 | 179 | 743
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.66 (10.08) | 54.69 (9.62) | 54.18 (10.14) | 54.76 (10.18) | 54.57 (9.98)
Age, Customized [Number; unit: participants]
  < 65 years | 159 | 159 | 155 | 153 | 626
  >= 65 years | 33 | 32 | 26 | 26 | 117
  >= 75 years | 3 | 2 | 5 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 88 | 86 | 83 | 366
  Male | 83 | 103 | 95 | 96 | 377
Race/Ethnicity, Customized [Number; unit: participants]
  White | 153 | 159 | 144 | 150 | 606
  Black / African American | 8 | 11 | 14 | 7 | 40
  Asian | 8 | 3 | 5 | 4 | 20
  Other | 23 | 18 | 18 | 18 | 77
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic / Latino | 27 | 25 | 29 | 27 | 108
  Not Hispanic / Latino | 64 | 62 | 54 | 49 | 229
  Not Reported | 101 | 104 | 98 | 103 | 406
Age Characterization Female Only [Number; unit: participants]
  =< 50 years | 33 | 34 | 24 | 21 | 112
  > 50 years | 76 | 54 | 62 | 62 | 254
Weight [Mean (Standard Deviation); unit: kg] | 85.97 (17.57) | 87.26 (17.04) | 87.83 (18.90) | 87.14 (17.75) | 87.04 (17.79)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.68 (5.15) | 31.23 (4.67) | 31.12 (4.79) | 31.57 (4.80) | 31.40 (4.85)
Body Mass Index Categorization [Number; unit: Participants]
  < 30 | 75 | 84 | 82 | 76 | 317
  >= 30 | 117 | 107 | 99 | 103 | 426

OUTCOME MEASURES:

1. Primary Outcome: Baseline and Change From Baseline in Hemoglobin A1c (A1C) at Week 24
Description: Mean change from baseline is adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized participants with both a baseline and post-baseline value (up to Week 24)
Measure: Mean (Standard Error); unit: percentage of glycosylated hemoglobins
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 186 | 186 | 180 | 175
percentage of glycosylated hemoglobins
  Baseline Mean | 8.08 (0.07) | 8.07 (0.06) | 7.98 (0.08) | 8.06 (0.07)
  Adjusted Mean Change from Baseline | -0.59 (0.07) | -0.69 (0.07) | -0.58 (0.07) | 0.13 (0.07)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, ANCOVA — Between-group comparisons significant at alpha = 0.019, significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-0.92 to -0.53], Standard Error of Mean 0.10 — ANCOVA model: difference between week t and baseline values = baseline values + treatment
Statistical Analysis 2: Comparison: Saxagliptin 5 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.02 to -0.63], Standard Error of Mean 0.10 — ANCOVA model: difference between week t and baseline values = baseline values + treatment
Statistical Analysis 3: Comparison: Saxagliptin 10 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF) .Adjusted for baseline; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-0.91 to -0.52], Standard Error of Mean 0.10 — ANCOVA model: difference between week t and baseline values = baseline values + treatment

2. Secondary Outcome: Baseline and Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Mean change from baseline is adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized Participants with measurement at timepoint. Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 188 | 187 | 181 | 176
mg/dL
  Baseline Mean | 173.57 (3.23) | 179.03 (3.44) | 175.86 (3.73) | 174.94 (3.27)
  Adjusted Mean Change from Baseline | -14.31 (2.48) | -22.03 (2.49) | -20.50 (2.53) | 1.24 (2.56)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -15.55, 95% CI 2-sided [-22.55 to -8.55], Standard Error of Mean 3.56 — ANCOVA model: difference between week t and baseline values = baseline values + treatment
Statistical Analysis 2: Comparison: Saxagliptin 5 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF) .Adjusted for baseline; Mean Difference (Final Values) = -23.28, 95% CI 2-sided [-30.29 to -16.27], Standard Error of Mean 3.57 — ANCOVA model: difference between week t and baseline values = baseline values + treatment
Statistical Analysis 3: Comparison: Saxagliptin 10 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF) .Adjusted for baseline; Mean Difference (Final Values) = -21.74, 95% CI 2-sided [-28.81 to -14.68], Standard Error of Mean 3.60 — ANCOVA model: difference between week t and baseline values = baseline values + treatment

3. Secondary Outcome: Percentage of Participants Achieving Therapeutic Glycemic Response (A1C < 7.0%) at Week 24
Time Frame: Week 24
Population: Randomized Participants with measurement at time point, Last Observation Carried Forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 186 | 186 | 180 | 175
percentage of participants | 37.1 | 43.5 | 44.4 | 16.6
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, Fisher Exact — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; The exact 95% CIs is based on the standardized statistic and inverting the one 2-sided test; Difference in Proportions = 20.5, 95% CI 2-sided [10.6 to 30.5]
Statistical Analysis 2: Comparison: Saxagliptin 5 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, Fisher Exact — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; The exact 95% CIs is based on the standardized statistic and inverting the one 2-sided test; Difference in Proportions = 27.0, 95% CI 2-sided [17.0 to 36.7]
Statistical Analysis 3: Comparison: Saxagliptin 10 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, Fisher Exact — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; The exact 95% CIs is based on the standardized statistic and inverting the one 2-sided test; Difference in Proportions = 27.9, 95% CI 2-sided [17.7 to 37.7]

4. Secondary Outcome: Baseline and Change From Baseline at Week 24 in Postprandial Glucose (PPG) Area Under the Curve (AUC)
Description: Mean change from baseline is adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized Participants with measurement at timepoint. Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 150 | 146 | 148 | 131
mg*min/dL
  Baseline Mean | 48224 (869.70) | 49021 (876.17) | 44931 (889.85) | 47407 (1071.9)
  Adjusted Mean Change from Baseline | -8891 (797.97) | -9586 (810.46) | -8137 (807.88) | -3291 (853.24)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -5599, 95% CI 2-sided [-7894 to -3305], Standard Error of Mean 1168.2 — ANCOVA model: difference between week t and baseline values = baseline values + treatment
Statistical Analysis 2: Comparison: Saxagliptin 5 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -6294, 95% CI 2-sided [-8606 to -3983], Standard Error of Mean 1176.8 — ANCOVA model: difference between week t and baseline values = baseline values + treatment
Statistical Analysis 3: Comparison: Saxagliptin 10 mg + Metformin vs Placebo+ Metformin; Test type: Superiority or Other; p < .0001, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -4845, 95% CI 2-sided [-7153 to -2537], Standard Error of Mean 1175.1 — ANCOVA model: difference between week t and baseline values = baseline values + treatment

5. Other Pre Specified Outcome: Overall Summary of Adverse Events During ST+LT Treatment Period
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event. Related events=relationship of certain, probable, possible, or missing.
Time Frame: AEs: up to last treatment day + 1 day or last visit day in the ST+LT period; SAEs: up to last treatment day + 30 days or last visit day + 30 days in the LT+ST period. Mean duration of exposure: 124, 118, 130, 95 wks respectively for 2.5mg, 5mg, 10 mg, pla
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
participants
  At Least 1 AE | 177 | 155 | 161 | 142
  At Least 1 Related AE | 53 | 57 | 65 | 56
  Deaths | 1 | 0 | 1 | 2
  At Least 1 SAE | 23 | 27 | 22 | 15
  At Least 1 Related SAE | 0 | 3 | 1 | 1
  Discontinuations Due to SAEs | 4 | 6 | 6 | 0
  Discontinuations Due to AEs | 11 | 18 | 13 | 9

6. Other Pre Specified Outcome: Marked Laboratory Abnormalities - During ST + LT Treatment Period
Description: A laboratory value was considered a marked abnormality if it is outside the pre-defined criteria for marked abnormality and the on-treatment value was more extreme (farther from the limit) than the baseline value. Pre-Rx=pretreatment; ULN=upper limit of normal; ALP=alkaline phosphatase; AST=aspartate aminotransferase; ALT=alanine aminotransferase; unspec=unspecified; sodium serum low: <0.9 x Pre-Rx & <=130mEq/L / high: >1.1 x Pre-Rx & >=150mEq/L; potassium, serum low: <=0.8 x Pre-Rx & >=6.0mEq/L / high: 1.2 x Pre-Rx & >=6.0mEq/L; LLN=lower limit of normal.
Time Frame: Lab assessments taken during and up to 14 days after the last dose of study drug during the ST + LT Treatment Period. Mean duration of exposure: 124, 118, 130, 95 weeks, respectively, for 2.5mg, 5mg, 10 mg, placebo.
Population: Number of Participants Analyzed=Treated participants; n=number of treated subjects with baseline value and at least one value during the ST + LT treatment period
Measure: Number; unit: participants
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
participants
  Hemoglobin < 8 g/dL (n=189, 190, 181, 179) | 1 | 1 | 1 | 0
  Hematocrit < 0.75 x pre-Rx (n=189, 190, 181, 179) | 2 | 5 | 5 | 2
  Platelets < 50 x 10^9 c/L (n=189, 188, 181, 178) | 0 | 0 | 0 | 0
  Platelets > 1.5 x ULN (n=189, 188, 181, 178) | 0 | 0 | 4 | 1
  Leukocytes < 2 x 1000 c/µL (n=189, 190, 181, 179) | 0 | 0 | 0 | 0
  Neutrophils+Bands <1x1000 c/µL (n=189,190,181,179) | 1 | 1 | 0 | 1
  Eosinophils >0.9x1000 c/µL (n=189, 190, 181, 179) | 12 | 12 | 18 | 9
  Lymphocytes <=0.75x1000 c/µL (n=189,190,181,179) | 3 | 4 | 4 | 2
  ALP >3 x pre-Rx and >ULN (n=190, 190, 181, 179) | 0 | 0 | 0 | 0
  ALP >1.5 x ULN (n=190, 190, 181, 179) | 3 | 1 | 1 | 3
  AST >3 x ULN (n=190, 190, 181, 179) | 6 | 1 | 3 | 0
  AST >5 x ULN (n=190, 190, 181, 179) | 1 | 0 | 1 | 0
  AST >10 x ULN (n=190, 190, 181, 179) | 0 | 0 | 0 | 0
  AST >20 x ULN (n=190, 190, 181, 179) | 0 | 0 | 0 | 0
  ALT >3 x ULN (n=190, 190, 181, 179) | 4 | 4 | 4 | 0
  ALT >5 x ULN (n=190, 190, 181, 179) | 1 | 0 | 1 | 0
  ALT >10 x ULN (n=190, 190, 181, 179) | 1 | 0 | 0 | 0
  ALT >20 x ULN (n=190, 190, 181, 179) | 0 | 0 | 0 | 0
  Bilirubin Total >2mg/dL (n=190,190,181,179) | 2 | 1 | 0 | 1
  Bilirubin Total >1.5xULN (n=190,190,181,179) | 2 | 1 | 0 | 1
  Bilirubin Total >2xULN (n=190,190,181,179) | 0 | 1 | 0 | 0
  BUN >2 x pre-Rx and >ULN (n=190,190,181,179) | 12 | 9 | 6 | 9
  Creatinine >2.5 mg/dL (n=190,190,181,179) | 1 | 1 | 1 | 1
  Glucose, Serum Fasting < 50 mg/dL (n=0, 0, 0, 0) | 0 | 0 | 0 | 0
  Glucose, Serum Fasting > 500 mg/dL (n=0, 0, 0, 0) | 0 | 0 | 0 | 0
  Glucose, Serum Unspec. < 50 mg/dL (n=0,0,0,0) | 0 | 0 | 0 | 0
  Glucose, Serum Unspec. > 500 mg/dL (n=0,0,0,0) | 0 | 0 | 0 | 0
  Glucose, Plasma Fasting<50mg/dL(n=189,189,181,179) | 2 | 3 | 1 | 3
  Glucose,Plasma Fasting>500mg/dL(n=189,189,181,179) | 0 | 0 | 0 | 0
  Glucose, Plasma Unspec.<50mg/dL(n=192,191,181,179) | 19 | 7 | 9 | 9
  Glucose,Plasma Unspec.>500mg/dL(n=192,191,181,179) | 1 | 1 | 1 | 1
  Sodium,Serum Low (*) (n=190,190,181,179) | 1 | 2 | 4 | 1
  Sodium,Serum High (*) (n=190,190,181,179) | 0 | 0 | 1 | 0
  Potassium, Serum Low (*) (n=190,190,181,179) | 0 | 1 | 1 | 1
  Potassium, Serum High (n=190,190,181,179) | 4 | 5 | 5 | 7
  Chloride < 90 mEq/L (n=190, 190, 181, 179) | 2 | 3 | 3 | 0
  Chloride > 120 mEq/L (n=190, 190, 181, 179) | 1 | 0 | 0 | 0
  Albumin < 0.9 LLN (n=190, 190, 181, 179) | 1 | 0 | 0 | 0
  Creatine Kinase > 5 x ULN (n=190, 190, 181, 179) | 1 | 2 | 3 | 1
  Uric Acid > 1.5 x ULN (n=0, 0, 0, 0) | 0 | 0 | 0 | 0
  Protein Urine, >=2-4 (n=187, 189, 180, 178) | 7 | 9 | 13 | 12
  Blood Urine, >=2-4 (n=187, 189, 180, 178) | 17 | 21 | 18 | 13
  Red Blood Cells Urine >=2-4 (n=175,176,162,166) | 28 | 27 | 22 | 20
  White Blood Cells Urine >=2-4 (n=175,176,162,166) | 43 | 38 | 26 | 28

7. Other Pre Specified Outcome: Baseline and Changes From Baseline in Hemoglobin During the ST + LT Period
Time Frame: Weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 30, 37, 50, 63, 76, 89, 102, 115, 128, 141, 154, 167, 180, 193, 206
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
g/dL
  Baseline (BL) (Week 0) (n=192, 191, 181, 179) | 14.06 (0.098) | 14.18 (0.094) | 14.18 (0.103) | 13.99 (0.096)
  Change from BL at Week 2 (n=181, 177, 172, 169) | -0.08 (0.044) | -0.18 (0.052) | -0.18 (0.044) | -0.09 (0.046)
  Change from BL at Week 4 (n=178, 178, 174, 166) | -0.07 (0.052) | -0.15 (0.047) | -0.09 (0.053) | 0.03 (0.056)
  Change from BL at Week 6 (n=176, 174, 166, 160) | -0.06 (0.052) | -0.15 (0.050) | -0.07 (0.050) | 0.00 (0.055)
  Change from BL at Week 8 (n=173, 176, 165, 157) | -0.07 (0.058) | -0.07 (0.051) | -0.02 (0.055) | 0.01 (0.056)
  Change from BL at Week 10 (n=149, 134, 137, 131) | -0.16 (0.061) | -0.17 (0.057) | -0.16 (0.067) | -0.16 (0.064)
  Change from BL at Week 12 (n=170, 167, 160, 144) | -0.05 (0.059) | -0.11 (0.054) | 0.03 (0.055) | -0.05 (0.065)
  Change from BL at Week 14 (n=156, 154, 146, 139) | -0.15 (0.059) | -0.20 (0.055) | -0.10 (0.068) | -0.02 (0.066)
  Change from BL at Week 16 (n=167, 166, 159, 140) | -0.12 (0.059) | -0.13 (0.052) | -0.10 (0.060) | -0.01 (0.060)
  Change from BL at Week 18 (n=155, 158, 149, 141) | -0.24 (0.069) | -0.28 (0.050) | -0.19 (0.059) | -0.09 (0.062)
  Change from BL at Week 20 (n=162, 153, 154, 147) | -0.16 (0.059) | -0.23 (0.061) | -0.10 (0.060) | -0.12 (0.060)
  Change from BL at Week 22 (n=157, 152, 143, 138) | -0.21 (0.064) | -0.33 (0.063) | -0.25 (0.062) | -0.23 (0.065)
  Change from BL at Week 24 (n=164, 160, 159, 137) | -0.23 (0.064) | -0.30 (0.063) | -0.25 (0.057) | -0.24 (0.065)
  Change from BL at Week 30 (n=161, 155, 154, 137) | -0.19 (0.059) | -0.29 (0.063) | -0.22 (0.071) | -0.18 (0.065)
  Change from BL at Week 37 (n=152, 149, 146, 122) | -0.17 (0.068) | -0.29 (0.064) | -0.19 (0.067) | -0.17 (0.066)
  Change from BL at Week 50 (n=151, 142, 146, 127) | -0.22 (0.061) | -0.22 (0.070) | -0.13 (0.066) | -0.12 (0.077)
  Change from BL at Week 63 (n=148, 137, 142, 116) | -0.10 (0.068) | -0.28 (0.096) | -0.17 (0.067) | -0.07 (0.073)
  Change from BL at Week 76 (n=134, 126, 130, 94) | -0.27 (0.077) | -0.31 (0.080) | -0.26 (0.066) | -0.26 (0.083)
  Change from BL at Week 89 (n=123, 114, 123, 85) | -0.22 (0.074) | -0.38 (0.075) | -0.32 (0.083) | -0.25 (0.088)
  Change from BL at Week 102 (n=108, 104, 112, 70) | -0.36 (0.073) | -0.40 (0.085) | -0.27 (0.078) | -0.34 (0.100)
  Change from BL at Week 115 (n=99, 94, 98, 58) | -0.26 (0.073) | -0.26 (0.082) | -0.36 (0.092) | -0.26 (0.106)
  Change from BL at Week 128 (n=92, 88, 90, 52) | -0.40 (0.095) | -0.41 (0.097) | -0.39 (0.095) | -0.28 (0.105)
  Change from BL at Week 141 (n=85, 79, 85, 48) | -0.49 (0.091) | -0.45 (0.093) | -0.42 (0.104) | -0.45 (0.132)
  Change from BL at Week 154 (n=81, 74, 78, 45) | -0.59 (0.092) | -0.56 (0.105) | -0.47 (0.102) | -0.57 (0.107)
  Change from BL at Week 167 (n=77, 67, 75, 42) | -0.49 (0.085) | -0.58 (0.127) | -0.53 (0.119) | -0.51 (0.137)
  Change from BL at Week 180 (n=70, 61, 73, 41) | -0.62 (0.099) | -0.81 (0.154) | -0.46 (0.107) | -0.53 (0.129)
  Change from BL at Week 193 (n=70, 60, 72, 40) | -0.60 (0.103) | -0.82 (0.159) | -0.47 (0.101) | -0.53 (0.134)
  Change from BL at Week 206 (n=61, 50, 64, 31) | -0.62 (0.108) | -0.87 (0.135) | -0.49 (0.101) | -0.75 (0.125)

8. Other Pre Specified Outcome: Baseline and Changes From Baseline in Hematocrit During the ST + LT Period
Time Frame: as for outcome 7
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: percentage red blood cells
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
percentage red blood cells
  Baseline (Week 0) (n=192, 191, 181, 179) | 41.9 (0.26) | 42.3 (0.25) | 42.2 (0.29) | 41.8 (0.28)
  Change from BL at Week 2 (n=181, 177, 172, 169) | -0.3 (0.15) | -0.5 (0.17) | -0.5 (0.15) | -0.4 (0.15)
  Change from BL at Week 4 (n=178, 178, 174, 166) | -0.3 (0.17) | -0.4 (0.15) | -0.2 (0.18) | -0.0 (0.17)
  Change from BL at Week 6 (n=176, 174, 166, 160) | -0.2 (0.17) | -0.3 (0.17) | -0.1 (0.18) | -0.0 (0.17)
  Change from BL at Week 8 (n=173, 176, 165, 157) | -0.4 (0.18) | -0.1 (0.17) | -0.0 (0.19) | -0.0 (0.19)
  Change from BL at Week 10 (n=149, 134, 137, 131) | -0.4 (0.19) | -0.4 (0.18) | -0.2 (0.21) | -0.1 (0.20)
  Change from BL at Week 12 (n=170, 167, 160, 144) | -0.1 (0.18) | -0.1 (0.17) | 0.4 (0.19) | 0.0 (0.20)
  Change from BL at Week 14 (n=156, 154, 146, 139) | -0.2 (0.18) | -0.2 (0.17) | -0.1 (0.23) | 0.0 (0.20)
  Change from BL at Week 16 (n=167, 166, 159, 140) | -0.1 (0.20) | 0.0 (0.18) | -0.1 (0.21) | 0.2 (0.19)
  Change from BL at Week 18 (n=155, 158, 149, 141) | -0.3 (0.21) | -0.5 (0.17) | -0.3 (0.18) | -0.1 (0.21)
  Change from BL at Week 20 (n=162, 153, 154, 147) | -0.1 (0.19) | -0.3 (0.19) | -0.2 (0.20) | -0.3 (0.20)
  Change from BL at Week 22 (n=157, 152, 143, 138) | -0.2 (0.21) | -0.5 (0.21) | -0.5 (0.21) | -0.5 (0.23)
  Change from BL at Week 24 (n=164, 160, 159, 137) | -0.3 (0.20) | -0.4 (0.21) | -0.3 (0.19) | -0.4 (0.22)
  Change from BL at Week 30 (n=161, 155, 154, 137) | -0.2 (0.19) | -0.4 (0.23) | -0.0 (0.21) | -0.2 (0.23)
  Change from BL at Week 37 (n=152, 149, 146, 122) | -0.1 (0.21) | -0.4 (0.21) | 0.0 (0.23) | -0.1 (0.21)
  Change from BL at Week 50 (n=151, 142, 146, 127) | -0.4 (0.21) | -0.5 (0.23) | -0.1 (0.22) | -0.0 (0.25)
  Change from BL at Week 63 (n=148, 137, 142, 116) | 0.1 (0.22) | -0.5 (0.28) | -0.1 (0.22) | -0.0 (0.24)
  Change from BL at Week 76 (n=134, 126, 130, 94) | -0.2 (0.25) | -0.4 (0.23) | 0.1 (0.22) | -0.4 (0.28)
  Change from BL at Week 89 (n=123, 114, 123, 85) | -0.2 (0.27) | -0.5 (0.25) | -0.3 (0.27) | -0.3 (0.29)
  Change from BL at Week 102 (n=108, 104, 112, 70) | -0.7 (0.21) | -0.9 (0.29) | -0.2 (0.25) | -0.7 (0.31)
  Change from BL at Week 115 (n=99, 94, 98, 58) | -0.1 (0.22) | 0.0 (0.29) | -0.4 (0.28) | -0.2 (0.33)
  Change from BL at Week 128 (n=92, 88, 90, 52) | -0.6 (0.27) | -0.5 (0.32) | -0.5 (0.28) | -0.5 (0.34)
  Change from BL at Week 141 (n=85, 79, 85, 48) | -0.6 (0.26) | -0.6 (0.28) | -0.3 (0.31) | -0.9 (0.37)
  Change from BL at Week 154 (n=81, 74, 78, 45) | -1.5 (0.28) | -1.7 (0.30) | -1.2 (0.32) | -1.6 (0.34)
  Change from BL at Week 167 (n=77, 67, 75, 42) | -1.0 (0.26) | -1.6 (0.34) | -1.2 (0.36) | -1.1 (0.41)
  Change from BL at Week 180 (n=70, 61, 73, 41) | -1.1 (0.32) | -1.8 (0.46) | -0.7 (0.30) | -1.2 (0.34)
  Change from BL at Week 193 (n=70, 60, 72, 40) | -0.7 (0.33) | -1.7 (0.46) | -0.5 (0.33) | -0.7 (0.42)
  Change from BL at Week 206 (n=61, 50, 64, 31) | -1.5 (0.35) | -2.3 (0.41) | -0.7 (0.32) | -1.3 (0.48)

9. Other Pre Specified Outcome: Baseline and Changes From Baseline in Red Blood Cell Counts (x 10^6 c/µL) During the ST + LT Period
Time Frame: as for outcome 7
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: 10^6 c/µL
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
10^6 c/µL
  Baseline (Week 0) (n=192, 191, 181, 179) | 4.68 (0.031) | 4.73 (0.029) | 4.70 (0.034) | 4.66 (0.033)
  Change from BL at Week 2 (n=181, 177, 172, 169) | -0.04 (0.015) | -0.05 (0.016) | -0.05 (0.015) | -0.03 (0.015)
  Change from BL at Week 4 (n=178, 178, 174, 166) | -0.02 (0.018) | -0.04 (0.016) | -0.01 (0.019) | 0.01 (0.018)
  Change from BL at Week 6 (n=176, 174, 166, 160) | -0.01 (0.017) | -0.02 (0.016) | 0.00 (0.018) | 0.03 (0.017)
  Change from BL at Week 8 (n=173, 176, 165, 157) | 0.00 (0.019) | 0.02 (0.017) | 0.03 (0.019) | 0.03 (0.019)
  Change from BL at Week 10 (n=149, 134, 137, 131) | -0.03 (0.020) | -0.02 (0.019) | 0.00 (0.021) | 0.00 (0.022)
  Change from BL at Week 12 (n=170, 167, 160, 144) | 0.03 (0.019) | 0.03 (0.018) | 0.09 (0.020) | 0.04 (0.022)
  Change from BL at Week 14 (n=156, 154, 146, 139) | 0.01 (0.019) | 0.01 (0.018) | 0.04 (0.024) | 0.04 (0.022)
  Change from BL at Week 16 (n=167, 166, 159, 140) | 0.04 (0.020) | 0.05 (0.017) | 0.07 (0.021) | 0.08 (0.020)
  Change from BL at Week 18 (n=155, 158, 149, 141) | 0.00 (0.024) | -0.01 (0.018) | 0.04 (0.018) | 0.03 (0.021)
  Change from BL at Week 20 (n=162, 153, 154, 147) | 0.02 (0.020) | 0.02 (0.020) | 0.06 (0.020) | 0.03 (0.021)
  Change from BL at Week 22 (n=157, 152, 143, 138) | 0.00 (0.022) | -0.03 (0.020) | 0.01 (0.020) | -0.02 (0.023)
  Change from BL at Week 24 (n=164, 160, 159, 137) | -0.02 (0.022) | -0.02 (0.020) | 0.01 (0.019) | -0.03 (0.024)
  Change from BL at Week 30 (n=161, 155, 154, 137) | -0.01 (0.020) | -0.02 (0.021) | 0.02 (0.022) | -0.01 (0.021)
  Change from BL at Week 37 (n=152, 149, 146, 122) | -0.00 (0.023) | -0.01 (0.019) | 0.02 (0.021) | 0.00 (0.022)
  Change from BL at Week 50 (n=151, 142, 146, 127) | -0.06 (0.022) | -0.04 (0.023) | 0.00 (0.021) | -0.03 (0.024)
  Change from BL at Week 63 (n=148, 137, 142, 116) | -0.01 (0.022) | -0.04 (0.031) | -0.01 (0.023) | -0.02 (0.024)
  Change from BL at Week 76 (n=134, 126, 130, 94) | -0.08 (0.025) | -0.06 (0.024) | -0.02 (0.023) | -0.09 (0.029)
  Change from BL at Week 89 (n=123, 114, 123, 85) | -0.09 (0.027) | -0.09 (0.024) | -0.07 (0.030) | -0.07 (0.028)
  Change from BL at Week 102 (n=108, 104, 112, 70) | -0.13 (0.024) | -0.12 (0.027) | -0.07 (0.027) | -0.14 (0.031)
  Change from BL at Week 115 (n=99, 94, 98, 58) | -0.08 (0.024) | -0.04 (0.026) | -0.06 (0.027) | -0.11 (0.034)
  Change from BL at Week 128 (n=92, 88, 90, 52) | -0.10 (0.028) | -0.07 (0.030) | -0.06 (0.027) | -0.08 (0.031)
  Change from BL at Week 141 (n=85, 79, 85, 48) | -0.13 (0.030) | -0.10 (0.027) | -0.06 (0.031) | -0.13 (0.041)
  Change from BL at Week 154 (n=81, 74, 78, 45) | -0.19 (0.032) | -0.17 (0.029) | -0.11 (0.029) | -0.20 (0.035)
  Change from BL at Week 167 (n=77, 67, 75, 42) | -0.14 (0.030) | -0.15 (0.032) | -0.12 (0.034) | -0.16 (0.041)
  Change from BL at Week 180 (n=70, 61, 73, 41) | -0.16 (0.033) | -0.21 (0.038) | -0.09 (0.033) | -0.16 (0.037)
  Change from BL at Week 193 (n=70, 60, 72, 40) | -0.14 (0.035) | -0.22 (0.040) | -0.12 (0.032) | -0.13 (0.044)
  Change from BL at Week 206 (n=61, 50, 64, 31) | -0.16 (0.040) | -0.25 (0.044) | -0.09 (0.032) | -0.15 (0.048)

10. Other Pre Specified Outcome: Baseline and Changes From Baseline in Platelet Counts (x 10^9 c/L) During the ST + LT Period
Time Frame: as for outcome 7
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: 10^9 c/L
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
10^9 c/L
  Baseline (Week 0) (n=192, 189, 181, 178) | 265.5 (4.78) | 256.2 (4.28) | 258.7 (5.05) | 261.0 (5.05)
  Change from BL at Week 2 (n=179, 168, 167, 166) | 8.4 (2.32) | 9.8 (2.77) | 6.5 (2.57) | 13.7 (2.99)
  Change from BL at Week 4 (n=176, 172, 168, 164) | 11.3 (2.59) | 11.8 (2.55) | 5.1 (2.31) | 11.1 (3.04)
  Change from BL at Week 6 (n=171, 171, 164, 157) | 8.7 (2.46) | 8.5 (2.78) | 5.1 (4.16) | 12.0 (2.99)
  Change from BL at Week 8 (n=172, 170, 162, 151) | 6.7 (2.53) | 7.5 (2.47) | 4.9 (2.67) | 8.5 (3.07)
  Change from BL at Week 10 (n=147, 132, 137, 129) | 4.7 (2.73) | 8.5 (3.23) | 0.5 (3.24) | 11.5 (3.30)
  Change from BL at Week 12 (n=170, 165, 157, 141) | 6.8 (2.49) | 9.3 (3.26) | 4.8 (3.24) | 8.2 (2.83)
  Change from BL at Week 14 (n=153, 149, 145, 133) | 6.1 (3.16) | 7.4 (2.70) | 2.5 (3.08) | 7.5 (2.70)
  Change from BL at Week 16 (n=166, 161, 156, 133) | 5.3 (2.71) | 7.1 (2.76) | -0.0 (2.64) | 7.4 (3.15)
  Change from BL at Week 18 (n=152, 155, 147, 139) | 5.6 (2.95) | 3.0 (2.66) | 5.2 (2.82) | 8.5 (3.59)
  Change from BL at Week 20 (n=160, 151, 153, 144) | 4.9 (3.00) | 7.0 (3.07) | -1.7 (2.64) | 6.8 (3.06)
  Change from BL at Week 22 (n=151, 148, 142, 134) | 3.5 (2.50) | 9.7 (2.98) | -1.7 (2.95) | 4.1 (3.24)
  Change from BL at Week 24 (n=158, 153, 156, 135) | 0.6 (2.97) | 3.5 (2.77) | -2.0 (2.75) | -2.3 (2.95)
  Change from BL at Week 30 (n=157, 153, 148, 130) | -0.1 (2.96) | 3.6 (2.88) | -0.8 (3.18) | 2.0 (3.65)
  Change from BL at Week 37 (n=149, 142, 139, 120) | -2.6 (3.07) | -4.1 (3.16) | -11.9 (2.98) | -2.3 (3.84)
  Change from BL at Week 50 (n=151, 141, 143, 120) | -3.2 (3.40) | -2.4 (3.44) | -9.0 (3.13) | -6.4 (3.70)
  Change from BL at Week 63 (n=147, 132, 137, 115) | 2.6 (3.24) | 3.5 (3.36) | 0.1 (4.80) | -4.7 (4.15)
  Change from BL at Week 76 (n=132, 124, 130, 92) | 0.1 (3.84) | 4.0 (3.55) | -2.6 (3.09) | 4.7 (3.98)
  Change from BL at Week 89 (n=122, 111, 122, 84) | 9.1 (4.42) | 8.6 (3.01) | 1.4 (3.68) | 13.6 (3.91)
  Change from BL at Week 102 (n=107, 103, 110, 69) | 0.3 (3.96) | 6.1 (3.47) | 3.3 (3.74) | 6.1 (5.20)
  Change from BL at Week 115 (n=99, 93, 98, 57) | 1.1 (4.45) | 4.2 (4.12) | 1.2 (4.19) | 7.0 (5.12)
  Change from BL at Week 128 (n=91, 84, 88, 51) | 5.7 (5.27) | 3.2 (3.89) | 2.2 (4.41) | 4.5 (4.73)
  Change from BL at Week 141 (n=83, 77, 84, 47) | 9.2 (4.96) | 6.5 (4.45) | 1.1 (5.21) | 12.0 (5.24)
  Change from BL at Week 154 (n=79, 70, 77, 45) | 8.0 (5.65) | 9.4 (4.55) | -1.8 (5.79) | 12.5 (7.01)
  Change from BL at Week 167 (n=75, 64, 74, 41) | 10.1 (5.39) | 3.2 (4.39) | -1.9 (5.26) | 13.8 (6.78)
  Change from BL at Week 180 (n=68, 60, 71, 41) | -2.7 (6.19) | -1.2 (5.65) | -8.3 (5.07) | 8.9 (5.80)
  Change from BL at Week 193 (n=67, 57, 68, 40) | 1.3 (6.40) | -2.9 (5.40) | -8.5 (5.19) | 12.2 (6.79)
  Change from BL at Week 206 (n=61, 49, 64, 31) | -0.7 (6.45) | 1.5 (7.48) | -4.7 (5.62) | 9.8 (7.45)

11. Other Pre Specified Outcome: Baseline and Changes From Baseline in White Blood Cell Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 7
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
10^3 c/µL
  Baseline (Week 0) (n=192, 191, 181, 179) | 7.23 (0.136) | 7.25 (0.167) | 7.12 (0.136) | 7.19 (0.136)
  Change from BL at Week 2 (n=178, 175, 171, 169) | 0.10 (0.093) | -0.03 (0.116) | 0.17 (0.102) | 0.11 (0.113)
  Change from BL at Week 4 (n=176, 176, 171, 166) | 0.19 (0.111) | 0.04 (0.131) | -0.02 (0.100) | 0.22 (0.117)
  Change from BL at Week 6 (n=175, 172, 165, 158) | 0.11 (0.089) | 0.02 (0.102) | 0.07 (0.092) | 0.07 (0.115)
  Change from BL at Week 8 (n=172, 174, 163, 153) | 0.15 (0.104) | -0.03 (0.116) | 0.19 (0.106) | 0.03 (0.109)
  Change from BL at Week 10 (n=148, 130, 137, 128) | 0.42 (0.108) | 0.37 (0.126) | 0.23 (0.105) | 0.39 (0.115)
  Change from BL at Week 12 (n=169, 166, 159, 142) | 0.18 (0.100) | 0.08 (0.134) | 0.26 (0.114) | 0.37 (0.130)
  Change from BL at Week 14 (n=156, 152, 145, 136) | 0.57 (0.142) | 0.30 (0.148) | 0.24 (0.121) | 0.33 (0.132)
  Change from BL at Week 16 (n=166, 166, 159, 137) | 0.28 (0.103) | 0.07 (0.127) | 0.16 (0.115) | 0.42 (0.139)
  Change from BL at Week 18 (n=155, 158, 149, 139) | 0.67 (0.121) | 0.23 (0.135) | 0.39 (0.114) | 0.58 (0.135)
  Change from BL at Week 20 (n=162, 153, 154, 146) | 0.23 (0.112) | -0.02 (0.130) | 0.19 (0.111) | 0.39 (0.142)
  Change from BL at Week 22 (n=157, 152, 143, 138) | 0.45 (0.112) | 0.36 (0.138) | 0.24 (0.112) | 0.50 (0.120)
  Change from BL at Week 24 (n=162, 160, 157, 135) | 0.13 (0.103) | 0.12 (0.161) | 0.11 (0.097) | 0.10 (0.135)
  Change from BL at Week 30 (n=160, 155, 154, 136) | 0.27 (0.091) | 0.05 (0.131) | 0.21 (0.109) | 0.14 (0.141)
  Change from BL at Week 37 (n=150, 149, 146, 121) | 0.34 (0.130) | 0.10 (0.137) | 0.02 (0.105) | 0.10 (0.135)
  Change from BL at Week 50 (n=150, 142, 145, 125) | -0.14 (0.116) | -0.14 (0.160) | -0.20 (0.114) | -0.36 (0.120)
  Change from BL at Week 63 (n=147, 136, 140, 115) | -0.10 (0.117) | -0.10 (0.123) | -0.02 (0.168) | -0.39 (0.148)
  Change from BL at Week 76 (n=134, 126, 130, 94) | -0.19 (0.122) | -0.18 (0.157) | -0.25 (0.105) | -0.30 (0.172)
  Change from BL at Week 89 (n=122, 114, 123, 85) | -0.29 (0.141) | -0.34 (0.136) | -0.21 (0.153) | -0.38 (0.197)
  Change from BL at Week 102 (n=105, 104, 111, 68) | -0.36 (0.140) | -0.11 (0.150) | -0.31 (0.102) | -0.54 (0.178)
  Change from BL at Week 115 (n=98, 92, 95, 57) | -0.10 (0.142) | -0.26 (0.161) | -0.05 (0.183) | -0.15 (0.202)
  Change from BL at Week 128 (n=90, 87, 88, 50) | -0.16 (0.162) | -0.27 (0.148) | -0.12 (0.155) | -0.32 (0.225)
  Change from BL at Week 141 (n=85, 78, 85, 47) | -0.01 (0.156) | -0.42 (0.161) | 0.13 (0.174) | -0.07 (0.235)
  Change from BL at Week 154 (n=77, 72, 78, 45) | -0.19 (0.170) | -0.38 (0.226) | -0.55 (0.144) | -0.54 (0.180)
  Change from BL at Week 167 (n=76, 67, 75, 42) | -0.15 (0.179) | -0.18 (0.178) | -0.18 (0.152) | -0.38 (0.177)
  Change from BL at Week 180 (n=70, 60, 72, 41) | -0.40 (0.185) | -0.72 (0.212) | -0.38 (0.142) | -0.37 (0.190)
  Change from BL at Week 193 (n=69, 60, 72, 40) | -0.45 (0.160) | -0.34 (0.228) | -0.13 (0.143) | -0.35 (0.203)
  Change from BL at Week 206 (n=61, 49, 63, 31) | -0.58 (0.175) | -0.80 (0.270) | -0.36 (0.170) | -0.71 (0.201)

12. Other Pre Specified Outcome: Baseline and Changes From Baseline in Absolute Neutrophil Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 7
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
10^3 c/µL
  Baseline (Week 0) (n=192, 191, 181, 179) | 4.27 (0.101) | 4.27 (0.127) | 4.19 (0.105) | 4.23 (0.102)
  Change from BL at Week 2 (n=178, 175, 170, 169) | 0.15 (0.083) | 0.05 (0.102) | 0.21 (0.087) | 0.12 (0.094)
  Change from BL at Week 4 (n=176, 175, 170, 166) | 0.21 (0.097) | 0.11 (0.116) | 0.15 (0.090) | 0.19 (0.098)
  Change from BL at Week 6 (n=175, 172, 165, 158) | 0.15 (0.075) | 0.10 (0.093) | 0.22 (0.085) | 0.07 (0.098)
  Change from BL at Week 8 (n=172, 172, 163, 153) | 0.16 (0.087) | 0.03 (0.103) | 0.35 (0.096) | 0.02 (0.097)
  Change from BL at Week 10 (n=148, 130, 137, 128) | 0.27 (0.094) | 0.28 (0.106) | 0.26 (0.093) | 0.19 (0.105)
  Change from BL at Week 12 (n=168, 166, 159, 141) | 0.22 (0.085) | 0.11 (0.110) | 0.40 (0.102) | 0.27 (0.111)
  Change from BL at Week 14 (n=156, 152, 145, 136) | 0.38 (0.123) | 0.24 (0.125) | 0.32 (0.109) | 0.17 (0.112)
  Change from BL at Week 16 (n=166, 166, 157, 137) | 0.24 (0.093) | 0.14 (0.113) | 0.30 (0.107) | 0.33 (0.113)
  Change from BL at Week 18 (n=155, 157, 149, 139) | 0.41 (0.104) | 0.16 (0.116) | 0.41 (0.099) | 0.34 (0.111)
  Change from BL at Week 20 (n=162, 153, 154, 146) | 0.17 (0.096) | 0.06 (0.109) | 0.32 (0.099) | 0.24 (0.122)
  Change from BL at Week 22 (n=157, 151, 143, 138) | 0.24 (0.096) | 0.24 (0.116) | 0.30 (0.097) | 0.24 (0.100)
  Change from BL at Week 24 (n=162, 160, 157, 135) | 0.06 (0.088) | 0.15 (0.150) | 0.20 (0.091) | 0.03 (0.111)
  Change from BL at Week 30 (n=159, 155, 154, 136) | 0.21 (0.085) | 0.03 (0.117) | 0.26 (0.090) | 0.04 (0.111)
  Change from BL at Week 37 (n=150, 149, 146, 121) | 0.27 (0.110) | 0.11 (0.122) | 0.20 (0.096) | 0.08 (0.105)
  Change from BL at Week 50 (n=150, 142, 145, 124) | -0.03 (0.104) | 0.02 (0.144) | -0.01 (0.107) | -0.25 (0.105)
  Change from BL at Week 63 (n=147, 136, 140, 115) | -0.05 (0.107) | 0.03 (0.100) | 0.23 (0.140) | -0.25 (0.119)
  Change from BL at Week 76 (n=134, 126, 130, 94) | -0.11 (0.108) | 0.02 (0.133) | 0.03 (0.101) | -0.13 (0.146)
  Change from BL at Week 89 (n=122, 113, 123, 85) | -0.17 (0.121) | -0.08 (0.106) | 0.08 (0.132) | -0.18 (0.163)
  Change from BL at Week 102 (n=104, 104, 111, 68) | -0.16 (0.123) | -0.04 (0.119) | -0.05 (0.093) | -0.35 (0.142)
  Change from BL at Week 115 (n=98, 92, 95, 57) | 0.00 (0.113) | -0.13 (0.145) | 0.11 (0.167) | -0.01 (0.169)
  Change from BL at Week 128 (n=90, 87, 88, 50) | -0.04 (0.147) | -0.04 (0.111) | 0.11 (0.136) | -0.11 (0.185)
  Change from BL at Week 141 (n=85, 78, 84, 47) | 0.00 (0.128) | -0.23 (0.131) | 0.32 (0.151) | 0.07 (0.195)
  Change from BL at Week 154 (n=77, 71, 78, 45) | 0.06 (0.167) | -0.10 (0.194) | -0.23 (0.117) | -0.34 (0.137)
  Change from BL at Week 167 (n=76, 67, 75, 42) | -0.04 (0.161) | 0.02 (0.160) | 0.06 (0.130) | -0.22 (0.145)
  Change from BL at Week 180 (n=69, 60, 72, 41) | -0.23 (0.159) | -0.35 (0.176) | -0.17 (0.114) | -0.20 (0.155)
  Change from BL at Week 193 (n=69, 60, 71, 40) | -0.25 (0.139) | -0.11 (0.178) | 0.11 (0.118) | -0.19 (0.185)
  Change from BL at Week 206 (n=61, 48, 63, 31) | -0.14 (0.146) | -0.40 (0.215) | -0.03 (0.124) | -0.29 (0.154)

13. Other Pre Specified Outcome: Baseline and Changes From Baseline in Absolute Lymphocyte Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 7
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
10^3 c/µL
  Baseline (Week 0) (n=192, 191, 181, 179) | 2.29 (0.051) | 2.29 (0.057) | 2.23 (0.051) | 2.31 (0.054)
  Change from BL at Week 2 (n=178, 175, 170, 169) | -0.02 (0.037) | -0.07 (0.036) | -0.03 (0.038) | -0.02 (0.038)
  Change from BL at Week 4 (n=176, 175, 170, 166) | -0.02 (0.035) | -0.04 (0.037) | -0.13 (0.035) | 0.00 (0.037)
  Change from BL at Week 6 (n=175, 172, 165, 158) | -0.03 (0.040) | -0.06 (0.033) | -0.12 (0.037) | -0.03 (0.038)
  Change from BL at Week 8 (n=172, 172, 163, 153) | -0.01 (0.038) | -0.04 (0.039) | -0.13 (0.038) | 0.00 (0.044)
  Change from BL at Week 10 (n=148, 130, 137, 128) | 0.12 (0.046) | 0.07 (0.049) | -0.03 (0.051) | 0.15 (0.046)
  Change from BL at Week 12 (n=168, 166, 159, 141) | -0.02 (0.041) | -0.02 (0.044) | -0.11 (0.043) | 0.07 (0.045)
  Change from BL at Week 14 (n=156, 152, 145, 136) | 0.13 (0.045) | 0.04 (0.039) | -0.08 (0.044) | 0.11 (0.048)
  Change from BL at Week 16 (n=166, 166, 157, 137) | 0.04 (0.045) | -0.08 (0.038) | -0.12 (0.047) | 0.04 (0.051)
  Change from BL at Week 18 (n=155, 157, 149, 139) | 0.22 (0.049) | 0.04 (0.044) | -0.06 (0.048) | 0.14 (0.050)
  Change from BL at Week 20 (n=162, 153, 154, 146) | 0.08 (0.040) | -0.07 (0.043) | -0.12 (0.039) | 0.10 (0.052)
  Change from BL at Week 22 (n=157, 151, 143, 138) | 0.16 (0.044) | 0.05 (0.043) | -0.09 (0.044) | 0.18 (0.047)
  Change from BL at Week 24 (n=162, 160, 157, 135) | 0.07 (0.045) | -0.02 (0.041) | -0.09 (0.039) | 0.02 (0.051)
  Change from BL at Week 30 (n=159, 155, 154, 136) | 0.06 (0.040) | 0.03 (0.045) | -0.07 (0.048) | 0.04 (0.051)
  Change from BL at Week 37 (n=150, 149, 146, 121) | 0.04 (0.045) | 0.00 (0.041) | -0.17 (0.048) | 0.00 (0.051)
  Change from BL at Week 50 (n=150, 142, 145, 124) | -0.12 (0.038) | -0.17 (0.040) | -0.25 (0.044) | -0.10 (0.042)
  Change from BL at Week 63 (n=147, 136, 140, 115) | -0.12 (0.042) | -0.17 (0.043) | -0.30 (0.042) | -0.16 (0.051)
  Change from BL at Week 76 (n=134, 126, 130, 94) | -0.11 (0.047) | -0.23 (0.044) | -0.30 (0.046) | -0.17 (0.054)
  Change from BL at Week 89 (n=122, 114, 123, 85) | -0.14 (0.053) | -0.23 (0.062) | -0.33 (0.047) | -0.21 (0.061)
  Change from BL at Week 102 (n=104, 104, 111, 68) | -0.20 (0.050) | -0.14 (0.058) | -0.30 (0.044) | -0.20 (0.063)
  Change from BL at Week 115 (n=98, 92, 95, 58) | -0.13 (0.057) | -0.15 (0.056) | -0.23 (0.057) | -0.12 (0.065)
  Change from BL at Week 128 (n=91, 88, 88, 50) | -0.15 (0.061) | -0.24 (0.057) | -0.28 (0.053) | -0.21 (0.075)
  Change from BL at Week 141 (n=85, 78, 84, 48) | -0.04 (0.067) | -0.20 (0.058) | -0.22 (0.060) | -0.17 (0.080)
  Change from BL at Week 154 (n=78, 71, 78, 45) | -0.23 (0.058) | -0.28 (0.079) | -0.35 (0.075) | -0.19 (0.065)
  Change from BL at Week 167 (n=77, 67, 75, 42) | -0.11 (0.065) | -0.25 (0.081) | -0.24 (0.058) | -0.13 (0.072)
  Change from BL at Week 180 (n=69, 60, 72, 41) | -0.21 (0.059) | -0.35 (0.072) | -0.26 (0.074) | -0.14 (0.081)
  Change from BL at Week 193 (n=69, 60, 71, 40) | -0.18 (0.069) | -0.31 (0.081) | -0.30 (0.071) | -0.14 (0.079)
  Change from BL at Week 206 (n=61, 48, 63, 31) | -0.40 (0.070) | -0.39 (0.085) | -0.36 (0.067) | -0.32 (0.077)

14. Other Pre Specified Outcome: Baseline and Changes From Baseline in Absolute Monocyte Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 7
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
10^3 c/µL
  Baseline (Week 0) (n=192, 191, 181, 179) | 0.40 (0.015) | 0.41 (0.015) | 0.42 (0.014) | 0.40 (0.014)
  Change from BL at Week 2 (n=178, 175, 170, 169) | -0.01 (0.015) | -0.01 (0.012) | -0.00 (0.011) | 0.01 (0.011)
  Change from BL at Week 4 (n=176, 175, 170, 166) | 0.01 (0.014) | -0.01 (0.014) | -0.01 (0.013) | 0.03 (0.012)
  Change from BL at Week 6 (n=175, 172, 165, 158) | 0.01 (0.013) | -0.01 (0.013) | 0.01 (0.011) | 0.02 (0.015)
  Change from BL at Week 8 (n=172, 172, 163, 153) | 0.00 (0.016) | -0.00 (0.013) | -0.02 (0.012) | 0.01 (0.013)
  Change from BL at Week 10 (n=148, 130, 137, 128) | 0.05 (0.016) | 0.02 (0.015) | 0.03 (0.012) | 0.05 (0.014)
  Change from BL at Week 12 (n=168, 166, 159, 141) | 0.02 (0.011) | 0.01 (0.013) | 0.01 (0.012) | 0.03 (0.014)
  Change from BL at Week 14 (n=156, 152, 145, 136) | 0.04 (0.015) | 0.03 (0.015) | 0.03 (0.014) | 0.05 (0.013)
  Change from BL at Week 16 (n=166, 166, 157, 137) | 0.02 (0.015) | 0.02 (0.014) | 0.02 (0.012) | 0.03 (0.014)
  Change from BL at Week 18 (n=155, 157, 149, 139) | 0.06 (0.015) | 0.04 (0.016) | 0.05 (0.014) | 0.06 (0.014)
  Change from BL at Week 20 (n=162, 153, 154, 146) | 0.02 (0.014) | 0.02 (0.014) | 0.02 (0.011) | 0.04 (0.012)
  Change from BL at Week 22 (n=157, 151, 143, 138) | 0.06 (0.015) | 0.04 (0.015) | 0.03 (0.012) | 0.07 (0.013)
  Change from BL at Week 24 (n=162, 160, 157, 135) | 0.03 (0.015) | 0.02 (0.015) | 0.02 (0.012) | 0.04 (0.013)
  Change from BL at Week 30 (n=159, 155, 154, 136) | 0.02 (0.013) | 0.02 (0.015) | 0.02 (0.011) | 0.05 (0.018)
  Change from BL at Week 37 (n=150, 149, 146, 121) | 0.03 (0.015) | 0.03 (0.017) | 0.02 (0.011) | 0.03 (0.016)
  Change from BL at Week 50 (n=150, 142, 145, 124) | 0.04 (0.014) | 0.04 (0.014) | 0.04 (0.011) | 0.03 (0.013)
  Change from BL at Week 63 (n=147, 136, 140, 115) | 0.06 (0.014) | 0.06 (0.016) | 0.06 (0.019) | 0.04 (0.015)
  Change from BL at Week 76 (n=134, 126, 130, 94) | 0.03 (0.015) | 0.05 (0.017) | 0.04 (0.012) | 0.05 (0.015)
  Change from BL at Week 89 (n=122, 113, 123, 85) | 0.04 (0.018) | 0.04 (0.019) | 0.06 (0.016) | 0.06 (0.017)
  Change from BL at Week 102 (n=104, 104, 111, 68) | 0.02 (0.018) | 0.07 (0.023) | 0.03 (0.015) | 0.06 (0.018)
  Change from BL at Week 115 (n=98, 92, 95, 57) | 0.04 (0.018) | 0.05 (0.023) | 0.08 (0.017) | 0.04 (0.019)
  Change from BL at Week 128 (n=90, 87, 88, 50) | 0.04 (0.021) | 0.05 (0.024) | 0.04 (0.014) | 0.04 (0.020)
  Change from BL at Week 141 (n=85, 78, 84, 47) | 0.05 (0.021) | 0.06 (0.021) | 0.07 (0.018) | 0.07 (0.019)
  Change from BL at Week 154 (n=77, 71, 78, 45) | 0.01 (0.021) | 0.07 (0.025) | 0.03 (0.019) | 0.05 (0.019)
  Change from BL at Week 167 (n=76, 67, 75, 42) | 0.01 (0.024) | 0.07 (0.024) | 0.03 (0.017) | 0.05 (0.017)
  Change from BL at Week 180 (n=69, 60, 72, 41) | 0.02 (0.024) | 0.04 (0.024) | 0.06 (0.017) | 0.04 (0.016)
  Change from BL at Week 193 (n=69, 60, 71, 40) | 0.01 (0.024) | 0.08 (0.027) | 0.06 (0.017) | 0.04 (0.014)
  Change from BL at Week 206 (n=61, 48, 63, 31) | 0.00 (0.018) | 0.04 (0.021) | 0.02 (0.019) | 0.01 (0.016)

15. Other Pre Specified Outcome: Baseline and Changes From Baseline in Absolute Basophil Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 7
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
10^3 c/µL
  Baseline (Week 0) (n=192, 191, 181, 179) | 0.02 (0.003) | 0.02 (0.003) | 0.02 (0.003) | 0.02 (0.003)
  Change from BL at Week 2 (n=178, 175, 170, 169) | -0.00 (0.002) | -0.00 (0.003) | 0.00 (0.003) | -0.00 (0.003)
  Change from BL at Week 4 (n=176, 175, 170, 166) | 0.00 (0.003) | -0.00 (0.003) | 0.00 (0.004) | -0.00 (0.003)
  Change from BL at Week 6 (n=175, 172, 165, 158) | -0.00 (0.003) | -0.00 (0.003) | -0.00 (0.003) | 0.00 (0.004)
  Change from BL at Week 8 (n=172, 172, 163, 153) | -0.00 (0.003) | -0.00 (0.003) | 0.00 (0.003) | -0.00 (0.003)
  Change from BL at Week 10 (n=148, 130, 137, 128) | -0.00 (0.003) | -0.00 (0.003) | -0.00 (0.003) | -0.00 (0.004)
  Change from BL at Week 12 (n=168, 166, 159, 141) | 0.00 (0.004) | 0.00 (0.004) | -0.00 (0.003) | -0.01 (0.003)
  Change from BL at Week 14 (n=156, 152, 145, 136) | -0.00 (0.003) | 0.00 (0.003) | -0.00 (0.003) | -0.01 (0.003)
  Change from BL at Week 16 (n=166, 166, 157, 137) | -0.00 (0.003) | 0.00 (0.003) | 0.00 (0.003) | -0.00 (0.003)
  Change from BL at Week 18 (n=155, 157, 149, 139) | 0.00 (0.004) | 0.00 (0.004) | 0.00 (0.003) | -0.00 (0.003)
  Change from BL at Week 20 (n=162, 153, 154, 146) | 0.00 (0.003) | -0.01 (0.003) | 0.00 (0.003) | -0.00 (0.004)
  Change from BL at Week 22 (n=157, 151, 143, 138) | 0.00 (0.003) | 0.00 (0.004) | -0.00 (0.003) | -0.00 (0.005)
  Change from BL at Week 24 (n=162, 160, 157, 135) | 0.00 (0.004) | 0.00 (0.003) | 0.00 (0.003) | -0.00 (0.004)
  Change from BL at Week 30 (n=159, 155, 154, 136) | 0.00 (0.003) | 0.00 (0.003) | 0.00 (0.004) | 0.00 (0.003)
  Change from BL at Week 37 (n=150, 149, 146, 121) | 0.00 (0.003) | 0.00 (0.003) | 0.01 (0.003) | -0.00 (0.004)
  Change from BL at Week 50 (n=150, 142, 145, 124) | 0.01 (0.003) | 0.01 (0.004) | 0.01 (0.003) | 0.00 (0.004)
  Change from BL at Week 63 (n=147, 136, 140, 115) | 0.01 (0.004) | 0.01 (0.004) | 0.01 (0.005) | 0.00 (0.004)
  Change from BL at Week 76 (n=134, 126, 130, 94) | 0.02 (0.005) | 0.01 (0.004) | 0.02 (0.005) | 0.00 (0.005)
  Change from BL at Week 89 (n=122, 113, 123, 85) | 0.01 (0.004) | 0.01 (0.004) | 0.01 (0.003) | 0.00 (0.005)
  Change from BL at Week 102 (n=104, 104, 111, 68) | 0.01 (0.005) | 0.01 (0.005) | 0.02 (0.005) | -0.00 (0.006)
  Change from BL at Week 115 (n=98, 92, 95, 57) | 0.01 (0.004) | 0.01 (0.006) | 0.01 (0.004) | 0.00 (0.007)
  Change from BL at Week 128 (n=90, 87, 88, 50) | 0.01 (0.005) | 0.01 (0.005) | 0.02 (0.005) | -0.00 (0.008)
  Change from BL at Week 141 (n=85, 78, 84, 47) | 0.01 (0.005) | 0.01 (0.004) | 0.01 (0.003) | -0.01 (0.008)
  Change from BL at Week 154 (n=77, 71, 78, 45) | 0.00 (0.005) | 0.01 (0.005) | 0.00 (0.005) | -0.01 (0.007)
  Change from BL at Week 167 (n=76, 67, 75, 42) | 0.01 (0.005) | 0.01 (0.006) | 0.01 (0.005) | -0.00 (0.008)
  Change from BL at Week 180 (n=69, 60, 72, 41) | -0.00 (0.005) | -0.00 (0.006) | 0.01 (0.004) | -0.01 (0.006)
  Change from BL at Week 193 (n=69, 60, 71, 40) | 0.01 (0.006) | 0.00 (0.006) | 0.00 (0.004) | -0.01 (0.008)
  Change from BL at Week 206 (n=61, 48, 63, 31) | 0.01 (0.005) | 0.01 (0.006) | 0.01 (0.005) | -0.01 (0.008)

16. Other Pre Specified Outcome: Baseline and Changes From Baseline in Absolute Eosinophil Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 7
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
10^3 c/µL
  Baseline (Week 0) (n=192, 191, 181, 179) | 0.24 (0.018) | 0.23 (0.016) | 0.24 (0.024) | 0.21 (0.013)
  Change from BL at Week 2 (n=178, 175, 170, 169) | -0.02 (0.014) | 0.01 (0.010) | -0.00 (0.013) | 0.00 (0.007)
  Change from BL at Week 4 (n=176, 175, 170, 166) | -0.01 (0.023) | -0.01 (0.011) | -0.02 (0.016) | 0.00 (0.007)
  Change from BL at Week 6 (n=175, 172, 165, 158) | -0.02 (0.017) | -0.01 (0.012) | -0.03 (0.012) | 0.01 (0.009)
  Change from BL at Week 8 (n=172, 172, 163, 153) | -0.00 (0.019) | -0.01 (0.011) | -0.02 (0.011) | 0.00 (0.010)
  Change from BL at Week 10 (n=148, 130, 137, 128) | -0.02 (0.012) | -0.01 (0.019) | -0.02 (0.015) | 0.01 (0.011)
  Change from BL at Week 12 (n=168, 166, 159, 141) | -0.02 (0.019) | -0.01 (0.013) | -0.03 (0.013) | 0.00 (0.009)
  Change from BL at Week 14 (n=156, 152, 145, 136) | 0.01 (0.022) | -0.01 (0.014) | -0.02 (0.016) | 0.02 (0.013)
  Change from BL at Week 16 (n=166, 166, 157, 137) | -0.02 (0.023) | 0.00 (0.012) | -0.02 (0.014) | 0.04 (0.016)
  Change from BL at Week 18 (n=155, 157, 149, 139) | -0.01 (0.015) | -0.00 (0.017) | -0.00 (0.013) | 0.04 (0.015)
  Change from BL at Week 20 (n=162, 153, 154, 146) | -0.04 (0.016) | -0.01 (0.014) | -0.02 (0.021) | 0.02 (0.013)
  Change from BL at Week 22 (n=157, 151, 143, 138) | -0.01 (0.017) | -0.00 (0.016) | 0.00 (0.011) | 0.03 (0.014)
  Change from BL at Week 24 (n=162, 160, 157, 135) | -0.03 (0.022) | -0.01 (0.021) | -0.01 (0.013) | 0.01 (0.011)
  Change from BL at Week 30 (n=159, 155, 154, 136) | -0.02 (0.017) | -0.01 (0.018) | 0.00 (0.012) | 0.00 (0.012)
  Change from BL at Week 37 (n=150, 149, 146, 121) | -0.00 (0.037) | -0.02 (0.016) | -0.03 (0.011) | -0.01 (0.011)
  Change from BL at Week 50 (n=150, 142, 145, 124) | -0.03 (0.021) | -0.02 (0.017) | 0.02 (0.030) | -0.02 (0.011)
  Change from BL at Week 63 (n=147, 136, 140, 115) | -0.00 (0.026) | -0.02 (0.018) | -0.01 (0.018) | -0.01 (0.015)
  Change from BL at Week 76 (n=134, 126, 130, 94) | -0.01 (0.031) | -0.01 (0.020) | -0.01 (0.014) | -0.03 (0.015)
  Change from BL at Week 89 (n=122, 113, 123, 85) | -0.02 (0.028) | -0.05 (0.023) | -0.01 (0.018) | -0.03 (0.015)
  Change from BL at Week 102 (n=104, 104, 111, 68) | -0.01 (0.052) | 0.00 (0.018) | 0.01 (0.015) | -0.03 (0.018)
  Change from BL at Week 115 (n=98, 92, 95, 57) | 0.00 (0.049) | -0.02 (0.025) | 0.00 (0.013) | -0.03 (0.022)
  Change from BL at Week 128 (n=90, 87, 88, 50) | -0.01 (0.051) | -0.02 (0.027) | 0.01 (0.015) | -0.03 (0.021)
  Change from BL at Week 141 (n=85, 78, 84, 47) | -0.01 (0.032) | -0.03 (0.024) | -0.01 (0.015) | -0.01 (0.032)
  Change from BL at Week 154 (n=77, 71, 78, 45) | -0.01 (0.051) | -0.02 (0.017) | -0.00 (0.018) | -0.03 (0.020)
  Change from BL at Week 167 (n=76, 67, 75, 42) | 0.01 (0.044) | -0.01 (0.014) | 0.00 (0.020) | -0.05 (0.019)
  Change from BL at Week 180 (n=69, 60, 72, 41) | 0.03 (0.044) | -0.03 (0.014) | -0.01 (0.017) | -0.04 (0.023)
  Change from BL at Week 193 (n=69, 60, 71, 40) | -0.02 (0.020) | -0.00 (0.021) | -0.00 (0.023) | -0.04 (0.025)
  Change from BL at Week 206 (n=61, 48, 63, 31) | -0.03 (0.019) | -0.03 (0.020) | 0.03 (0.031) | -0.09 (0.028)

17. Other Pre Specified Outcome: Changes From Baseline in Systolic Blood Pressure During the ST + LT Period
Time Frame: Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 30, 37, 50, 63, 76, 89, 102, 115, 128, 141, 154, 167, 180, 193, 206
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
mmHg
  Change from BL at Week 2 (n=182, 181, 176, 170) | -1.6 (1.0) | -2.5 (1.0) | -1.6 (0.9) | -3.3 (1.1)
  Change from BL at Week 4 (n=178, 179, 175, 164) | -2.0 (1.0) | -2.3 (1.1) | -3.3 (0.9) | -2.9 (1.1)
  Change from BL at Week 6 (n=178, 176, 171, 162) | -2.8 (1.1) | -4.1 (1.0) | -2.8 (1.1) | -2.8 (1.1)
  Change from BL at Week 8 (n=175, 176, 170, 152) | -2.9 (1.1) | -4.2 (1.1) | -4.2 (1.1) | -3.7 (1.2)
  Change from BL at Week 10 (n=116, 108, 101, 101) | -2.1 (1.4) | -3.3 (1.2) | -2.8 (1.4) | -6.8 (1.5)
  Change from BL at Week 12 (n=170, 166, 161, 138) | -2.2 (1.1) | -2.8 (1.1) | -4.3 (1.0) | -4.3 (1.3)
  Change from BL at Week 14 (n=132, 129, 124, 116) | -0.7 (1.3) | -2.3 (1.1) | -3.4 (1.1) | -2.6 (1.4)
  Change from BL at Week 16 (n=166, 164, 156, 140) | -2.7 (1.1) | -3.5 (1.1) | -4.4 (1.0) | -2.6 (1.2)
  Change from BL at Week 18 (n=144, 141, 132, 123) | -1.9 (1.2) | -2.2 (1.2) | -4.2 (1.1) | -4.1 (1.4)
  Change from BL at Week 20 (n=163, 155, 153, 147) | -2.9 (1.2) | -2.2 (1.1) | -4.9 (1.2) | -4.3 (1.3)
  Change from BL at Week 22 (n=146, 140, 136, 126) | -2.0 (1.2) | -3.1 (1.2) | -3.1 (1.2) | -4.7 (1.3)
  Change from BL at Week 24 (n=165, 160, 161, 140) | -4.3 (1.2) | -3.6 (1.2) | -3.8 (1.2) | -4.5 (1.3)
  Change from BL at Week 30 (n=162, 156, 155, 138) | -3.6 (1.2) | -1.1 (1.3) | -2.5 (1.2) | -3.4 (1.4)
  Change from BL at Week 37 (n=154, 151, 149, 123) | -2.6 (1.2) | -1.8 (1.3) | -3.3 (1.3) | -2.3 (1.2)
  Change from BL at Week 50 (n=155, 147, 151, 130) | -2.6 (1.3) | -1.7 (1.2) | -1.9 (1.2) | -2.9 (1.5)
  Change from BL at Week 63 (n=151, 138, 145, 117) | -0.6 (1.3) | 0.9 (1.2) | -0.6 (1.3) | -0.0 (1.3)
  Change from BL at Week 76 (n=134, 126, 133, 98) | -0.1 (1.5) | -0.6 (1.4) | -0.7 (1.3) | -1.7 (1.6)
  Change from BL at Week 89 (n=124, 117, 125, 86) | -3.7 (1.3) | 0.3 (1.4) | -1.7 (1.4) | 0.3 (1.6)
  Change from BL at Week 102 (n=111, 107, 113, 73) | -3.2 (1.5) | 0.6 (1.5) | -2.8 (1.4) | -2.0 (2.0)
  Change from BL at Week 115 (n=100, 94, 98, 58) | -0.4 (1.8) | 2.0 (1.8) | -1.3 (1.6) | -2.8 (1.9)
  Change from BL at Week 128 (n=94, 88, 90, 52) | -0.4 (1.7) | 2.9 (2.0) | 1.5 (1.7) | -2.5 (2.0)
  Change from BL at Week 141 (n=87, 82, 85, 49) | -0.7 (1.8) | 2.0 (1.6) | -1.5 (1.7) | 0.3 (2.3)
  Change from BL at Week 154 (n=84, 75, 79, 45) | 0.3 (1.7) | -0.0 (1.8) | 1.5 (1.8) | -2.8 (2.3)
  Change from BL at Week 167 (n=78, 67, 75, 42) | 0.8 (1.7) | -0.4 (2.1) | 0.7 (1.7) | -1.8 (2.5)
  Change from BL at Week 180 (n=71, 63, 74, 41) | -0.0 (2.0) | 3.1 (2.1) | 3.5 (1.7) | 2.7 (2.5)
  Change from BL at Week 193 (n=70, 60, 72, 40) | -0.1 (2.0) | 0.9 (2.3) | 0.2 (1.8) | -1.4 (2.4)
  Change from BL at Week 206 (n=61, 53, 64, 33) | -2.6 (2.1) | 2.2 (2.3) | 1.7 (1.9) | -0.4 (2.2)

18. Other Pre Specified Outcome: Changes From Baseline in Diastolic Blood Pressure During the ST + LT Period
Time Frame: Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 30, 37, 50, 63, 76, 89, 102, 115, 128, 141, 154, 167, 180, 193, 206
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
mmHg
  Change from BL at Week 2 (n=182, 181, 176, 170) | -1.0 (0.6) | -1.1 (0.7) | -0.9 (0.6) | -1.5 (0.7)
  Change from BL at Week 4 (n=178, 179, 175, 164) | -0.3 (0.7) | -0.9 (0.7) | -1.3 (0.6) | -1.4 (0.7)
  Change from BL at Week 6 (n=178, 176, 171, 162) | -0.1 (0.7) | -1.6 (0.7) | -0.5 (0.6) | -1.4 (0.7)
  Change from BL at Week 8 (n=175, 176, 170, 152) | -1.1 (0.7) | -1.9 (0.7) | -1.5 (0.6) | -2.2 (0.7)
  Change from BL at Week 10 (n=116, 108, 101, 101) | 0.3 (0.8) | -0.5 (0.8) | -1.6 (0.8) | -3.4 (0.9)
  Change from BL at Week 12 (n=170, 166, 161, 138) | -0.6 (0.7) | -1.0 (0.7) | -2.1 (0.6) | -1.7 (0.8)
  Change from BL at Week 14 (n=132, 129, 124, 116) | -0.2 (0.8) | -0.4 (0.7) | -2.2 (0.7) | -2.1 (0.9)
  Change from BL at Week 16 (n=166, 164, 156, 140) | -0.7 (0.7) | -1.0 (0.6) | -1.7 (0.6) | -1.0 (0.8)
  Change from BL at Week 18 (n=144, 141, 132, 123) | -1.4 (0.8) | -0.7 (0.8) | -2.3 (0.7) | -1.8 (0.8)
  Change from BL at Week 20 (n=163, 155, 153, 147) | -1.2 (0.7) | -1.0 (0.7) | -2.1 (0.7) | -1.9 (0.7)
  Change from BL at Week 22 (n=146, 140, 136, 126) | -0.7 (0.8) | -1.2 (0.8) | -1.6 (0.8) | -1.6 (0.8)
  Change from BL at Week 24 (n=165, 160, 161, 140) | -1.3 (0.7) | -1.3 (0.8) | -2.5 (0.7) | -2.4 (0.7)
  Change from BL at Week 30 (n=162, 156, 155, 138) | -0.9 (0.8) | -0.5 (0.8) | -1.6 (0.7) | -1.6 (0.8)
  Change from BL at Week 37 (n=154, 151, 149, 123) | -0.9 (0.7) | -1.1 (0.8) | -1.9 (0.8) | -1.6 (0.8)
  Change from BL at Week 50 (n=155, 147, 151, 130) | -1.1 (0.8) | -1.7 (0.8) | -1.5 (0.7) | -1.4 (0.8)
  Change from BL at Week 63 (n=151, 138, 145, 117) | -0.8 (0.8) | -0.3 (0.7) | -0.9 (0.7) | -0.7 (0.8)
  Change from BL at Week 76 (n=134, 126, 133, 98) | -0.2 (0.9) | -1.2 (0.8) | -1.6 (0.8) | -1.8 (1.0)
  Change from BL at Week 89 (n=124, 117, 125, 86) | -1.2 (0.8) | -0.8 (0.8) | -1.9 (0.8) | -2.1 (1.0)
  Change from BL at Week 102 (n=111, 107, 113, 73) | -2.2 (0.9) | -0.4 (1.0) | -2.3 (0.9) | -3.6 (1.2)
  Change from BL at Week 115 (n=100, 94, 98, 58) | -0.1 (1.0) | 0.7 (1.1) | -1.1 (1.1) | -3.6 (1.2)
  Change from BL at Week 128 (n=94, 88, 90, 52) | -0.6 (1.1) | 0.0 (1.1) | -1.2 (1.0) | -3.1 (1.3)
  Change from BL at Week 141 (n=87, 82, 85, 49) | 0.7 (1.1) | 0.3 (1.1) | -3.0 (1.1) | -2.7 (1.5)
  Change from BL at Week 154 (n=84, 75, 79, 45) | -0.7 (1.0) | -1.8 (1.1) | -2.7 (1.1) | -4.6 (1.2)
  Change from BL at Week 167 (n=78, 67, 75, 42) | 2.1 (1.0) | -1.4 (1.3) | -1.6 (1.2) | -2.0 (1.7)
  Change from BL at Week 180 (n=71, 63, 74, 41) | -0.3 (0.9) | -1.4 (1.2) | -0.9 (1.2) | -1.6 (1.7)
  Change from BL at Week 193 (n=70, 60, 72, 40) | 0.4 (1.2) | -2.6 (1.3) | -1.7 (1.2) | -2.6 (1.6)
  Change from BL at Week 206 (n=61, 53, 64, 33) | -2.8 (1.0) | -0.6 (1.4) | -2.3 (1.3) | -2.8 (1.6)

19. Other Pre Specified Outcome: Changes From Baseline in Heart Rate During the ST + LT Period
Time Frame: Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 30, 37, 50, 63, 76, 89, 102, 115, 128, 141, 154, 167, 180, 193, 206
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: beats/min
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
beats/min
  Change from BL at Week 2 (n=182, 181, 176, 170) | -0.3 (0.7) | 1.0 (0.7) | -0.4 (0.8) | 0.7 (0.7)
  Change from BL at Week 4 (n=178, 179, 175, 164) | -0.1 (0.8) | 1.3 (0.6) | -0.0 (0.7) | 0.1 (0.6)
  Change from BL at Week 6 (n=178, 176, 171, 162) | -0.2 (0.7) | 1.0 (0.6) | -0.2 (0.7) | -0.5 (0.7)
  Change from BL at Week 8 (n=175, 176, 170, 152) | 0.5 (0.7) | 0.8 (0.6) | 0.6 (0.7) | -0.6 (0.7)
  Change from BL at Week 10 (n=116, 106, 100, 101) | -0.5 (0.8) | 0.9 (0.8) | 0.2 (1.0) | -1.5 (0.9)
  Change from BL at Week 12 (n=170, 166, 161, 138) | -0.2 (0.7) | 0.7 (0.6) | 0.1 (0.7) | -1.5 (0.8)
  Change from BL at Week 14 (n=132, 129, 124, 116) | -0.1 (0.8) | 1.4 (0.8) | 1.0 (0.9) | -1.5 (0.9)
  Change from BL at Week 16 (n=166, 164, 156, 140) | -0.6 (0.7) | 0.4 (0.7) | -0.5 (0.8) | -0.5 (0.8)
  Change from BL at Week 18 (n=144, 141, 132, 123) | -0.0 (0.8) | 1.6 (0.8) | 0.3 (0.8) | -0.5 (0.9)
  Change from BL at Week 20 (n=163, 155, 153, 147) | -0.0 (0.7) | 0.9 (0.7) | -0.3 (0.8) | -0.8 (0.8)
  Change from BL at Week 22 (n=146, 140, 136, 126) | 0.4 (0.9) | 2.4 (0.8) | 0.3 (0.8) | -1.6 (0.9)
  Change from BL at Week 24 (n=165, 160, 161, 140) | -0.6 (0.8) | 0.2 (0.7) | 0.4 (0.7) | -0.7 (0.7)
  Change from BL at Week 30 (n=162, 156, 154, 138) | -0.7 (0.8) | 0.5 (0.7) | -0.3 (0.8) | -0.1 (0.8)
  Change from BL at Week 37 (n=154, 151, 149, 123) | -1.2 (0.8) | 0.6 (0.7) | -0.3 (0.8) | -0.6 (0.8)
  Change from BL at Week 50 (n=154, 147, 151, 130) | -1.0 (0.8) | 0.8 (0.8) | 0.1 (0.8) | -1.0 (0.8)
  Change from BL at Week 63 (n=151, 138, 145, 117) | -0.8 (0.8) | 0.4 (0.8) | -0.8 (0.7) | -0.5 (0.9)
  Change from BL at Week 76 (n=134, 126, 133, 98) | -1.3 (0.8) | -0.0 (0.9) | -0.5 (0.9) | -1.4 (0.9)
  Change from BL at Week 89 (n=124, 116, 125, 86) | -1.5 (0.8) | -0.3 (0.9) | -0.2 (0.8) | -1.6 (1.0)
  Change from BL at Week 102 (n=111, 107, 113, 73) | -0.6 (0.9) | 0.5 (0.9) | 0.6 (0.8) | -1.8 (1.2)
  Change from BL at Week 115 (n=100, 94, 98, 58) | -0.5 (0.9) | -0.3 (1.1) | -0.8 (1.0) | -2.4 (1.2)
  Change from BL at Week 128 (n=94, 88, 90, 52) | -0.2 (0.9) | -0.7 (1.2) | -0.9 (1.1) | -0.9 (1.3)
  Change from BL at Week 141 (n=87, 82, 85, 49) | -1.7 (1.0) | -1.7 (1.2) | -0.6 (1.2) | -1.2 (1.3)
  Change from BL at Week 154 (n=84, 75, 79, 45) | -0.6 (0.9) | -0.9 (1.4) | -0.0 (1.2) | -2.8 (1.4)
  Change from BL at Week 167 (n=78, 67, 75, 42) | 0.3 (1.0) | -0.0 (1.3) | -1.2 (1.2) | -0.9 (1.4)
  Change from BL at Week 180 (n=71, 63, 74, 41) | -0.8 (1.1) | -2.8 (1.3) | 0.2 (1.6) | -2.7 (1.3)
  Change from BL at Week 193 (n=70, 60, 72, 40) | -0.3 (1.1) | -2.2 (1.3) | -1.1 (1.1) | -1.8 (1.5)
  Change from BL at Week 206 (n=61, 53, 64, 33) | 0.1 (1.2) | -0.9 (1.2) | -1.2 (1.2) | -1.1 (1.6)

20. Other Pre Specified Outcome: Electrocardiogram (ECG) Tracings - Shift Table From Baseline (BL) to Selected Visits During ST + LT Treatment Period
Description: The normality/abnormality of the ECG tracing was determined by the investigator.
Time Frame: Baseline, Weeks 12, 24, 76, 102, 154, 206,
Population: Number of Participants Analyzed=Treated Participants; BL n=normal or abnormal ECG status at baseline of the cohort of participants with measure at given time point
Measure: Number; unit: participants
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
participants
  Normal BL, Normal Week 12(BL n=108, 109, 104, 104) | 97 | 98 | 94 | 82
  Normal BL, Abnormal Week 12 (BL n=108,109,104,104) | 11 | 11 | 10 | 22
  Abnormal BL, Normal Week 12 (BL n=69, 66, 70, 58) | 14 | 22 | 22 | 12
  Abnormal BL, Abnormal Week 12(BL n=69, 66, 70, 58) | 55 | 44 | 48 | 46
  Normal BL, Normal Week 24 (BL n=96, 87, 83, 77) | 82 | 79 | 70 | 61
  Normal BL, Abnormal Week 24 (BL n=96, 87, 83, 77) | 14 | 8 | 13 | 16
  Abnormal BL, Normal Week 24 (BL n=58, 58, 56, 41) | 16 | 22 | 15 | 14
  Abnormal BL, Abnormal Week 24(BL n=58, 58, 56, 41) | 42 | 36 | 41 | 27
  Normal BL, Normal Week 76 (BL n=94, 89, 92, 81) | 75 | 74 | 73 | 60
  Normal BL, Abnormal Week 76 (BL n=94, 89, 92, 81) | 19 | 15 | 19 | 21
  Abnormal BL, Normal Week 76 (BL n=51, 52, 59, 44) | 13 | 18 | 18 | 13
  Abnormal BL, Abnormal Week 76 (BL n=51,52,59,44) | 38 | 34 | 41 | 31
  Normal BL, Normal Week 102 (BL n=80, 66, 65, 50) | 63 | 55 | 48 | 41
  Normal BL, Abnormal Week 102 (BL n=80, 66, 65, 50) | 17 | 11 | 17 | 9
  Abnormal BL, Normal Week 102 (BL n=43,45,49, 21) | 11 | 14 | 14 | 6
  Abnormal BL, Abnormal Week 102 (BL n=43,45,49, 21) | 32 | 31 | 35 | 15
  Normal BL, Normal Week 154 (BL n=60, 46, 53, 34) | 48 | 36 | 37 | 26
  Normal BL, Abnormal Week 154 (BL n=60, 46, 53, 34) | 12 | 10 | 16 | 8
  Abnormal BL, Normal Week 154 (BL n=26, 34, 34, 16) | 10 | 13 | 12 | 7
  Abnormal BL, Abnormal Week 154 (BL n=26,34,34,16) | 16 | 21 | 22 | 9
  Normal BL, Normal Week 206 (BL n=48, 31, 42, 24) | 39 | 27 | 32 | 16
  Normal BL, Abnormal Week 206 (BL n=48, 31, 42, 24) | 9 | 4 | 10 | 8
  Abnormal BL, Normal Week 206 (BL n=20, 25, 28, 13) | 9 | 9 | 11 | 7
  Abnormal BL, Abnormal Week 206 (BL n=20,25,28,13) | 11 | 16 | 17 | 6

21. Other Pre Specified Outcome: All Reported Hypoglycemic Adverse Events During the ST + LT Treatment Period
Description: Hypoglycemic Events are based upon the Saxagliptin Predefined List of Events, which are hypoglycemia, blood glucose decreased, and hypoglycemic unconsciousness.
Time Frame: as for outcome 5
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
participants | 23 | 20 | 21 | 20

22. Other Pre Specified Outcome: Confirmed Hypoglycemia During the ST + LT Treatment Period
Description: 'Confirmed' = recorded on the hypoglycemia AE case report form with a fingerstick glucose <= 50 mg/dL and associated symptoms.
Time Frame: as for outcome 5
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Placebo+ Metformin
Number analyzed (Participants) | 192 | 191 | 181 | 179
participants | 3 | 2 | 3 | 1

ADVERSE EVENTS:
Arm/Group | Placebo+ Metformin | Saxagliptin 10 mg + Metformin | Saxagliptin 2.5 mg + Metformin | Saxagliptin 5 mg + Metformin
Serious Adverse Events (participants affected / at risk) | 15/179 | 22/181 | 23/192 | 27/191
Other Adverse Events (participants affected / at risk) | 129/179 | 133/181 | 139/192 | 133/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+ Metformin (N=179) | Saxagliptin 10 mg + Metformin (N=181) | Saxagliptin 2.5 mg + Metformin (N=192) | Saxagliptin 5 mg + Metformin (N=191)
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0 | 0 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 0 | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 2 | 0 | 4
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 0 | 0 | 3
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0 | 0
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 0 | 0 | 1 | 0
VARICOSE VEIN (Vascular disorders) | 0 | 0 | 0 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 1 | 1 | 0 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 1 | 0 | 1 | 0
PSYCHIATRIC SYMPTOM (Psychiatric disorders) | 0 | 1 | 0 | 0
BILIARY COLIC (Hepatobiliary disorders) | 0 | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 1 | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 1 | 0
SARCOIDOSIS (Immune system disorders) | 0 | 0 | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 3 | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 0 | 0 | 1
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1
FOOD POISONING (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 1 | 0
STOMACH GRANULOMA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 2 | 1
SINUSITIS (Infections and infestations) | 0 | 1 | 0 | 0
UROSEPSIS (Infections and infestations) | 0 | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 0 | 1 | 0
BREAST ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 1 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 1 | 0 | 0
SCROTAL ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
SINUSITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 0
PERIUMBILICAL ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
MENINGITIS TUBERCULOUS (Infections and infestations) | 0 | 1 | 0 | 0
APPENDICITIS PERFORATED (Infections and infestations) | 0 | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 1 | 0 | 1
CALCULUS URINARY (Renal and urinary disorders) | 0 | 0 | 0 | 1
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 1 | 0
STERILISATION (Surgical and medical procedures) | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
CYSTOCELE (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
RECTOCELE (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
DYSFUNCTIONAL UTERINE BLEEDING (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
HERNIA (General disorders) | 0 | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 1 | 0
PELVIC MASS (General disorders) | 0 | 1 | 0 | 0
NEURILEMMOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
BREAST CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+ Metformin (N=179) | Saxagliptin 10 mg + Metformin (N=181) | Saxagliptin 2.5 mg + Metformin (N=192) | Saxagliptin 5 mg + Metformin (N=191)
HYPERTENSION (Vascular disorders) | 13 | 16 | 21 | 14
HEADACHE (Nervous system disorders) | 22 | 24 | 27 | 18
DIZZINESS (Nervous system disorders) | 10 | 8 | 9 | 8
NAUSEA (Gastrointestinal disorders) | 8 | 14 | 11 | 7
VOMITING (Gastrointestinal disorders) | 8 | 7 | 12 | 9
DIARRHOEA (Gastrointestinal disorders) | 23 | 19 | 29 | 19
DYSPEPSIA (Gastrointestinal disorders) | 8 | 6 | 9 | 12
GASTRITIS (Gastrointestinal disorders) | 2 | 4 | 10 | 3
TOOTHACHE (Gastrointestinal disorders) | 11 | 2 | 6 | 10
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 5 | 13 | 8
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 | 6 | 6 | 10
INFLUENZA (Infections and infestations) | 27 | 28 | 27 | 31
SINUSITIS (Infections and infestations) | 8 | 15 | 9 | 14
BRONCHITIS (Infections and infestations) | 13 | 12 | 15 | 19
GASTROENTERITIS (Infections and infestations) | 4 | 5 | 10 | 6
NASOPHARYNGITIS (Infections and infestations) | 25 | 28 | 28 | 28
URINARY TRACT INFECTION (Infections and infestations) | 15 | 22 | 26 | 16
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 17 | 21 | 25 | 19
ANAEMIA (Blood and lymphatic system disorders) | 4 | 5 | 7 | 15
RASH (Skin and subcutaneous tissue disorders) | 5 | 12 | 5 | 6
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 8 | 10 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 19 | 14 | 19 | 16
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 | 23 | 22 | 20
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 17 | 15 | 14 | 10
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 9 | 10 | 5 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 15 | 9
OEDEMA PERIPHERAL (General disorders) | 12 | 16 | 16 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.